CLINICAL TRIAL: NCT05429021
Title: A Randomized, Double-Blind, Placebo-Controlled, First-in-Human, Phase 1 Study to Evaluate the Safety, Pharmacokinetics, and Viral Clearance of Single Ascending Doses of IMM-BCP-01 Administered Intravenously in Adults With Mild to Moderate COVID-19
Brief Title: IMM-BCP-01 in Mild to Moderate COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision to discontinue the study based on strategic prioritization.
Sponsor: Immunome, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: IMM-BCP-1001
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: SARS-CoV2 Infection; COVID-19
Keywords: IMM-BCP-01; antibody cocktail
MeSH Terms: conditions — COVID-19 | interventions — IMM20184, IMM20190, and IMM20253 drug combination

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Dose Escalation
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IV Cohort 1 (Experimental): Single intravenous (IV) dose 1 of IMM-BCP-01 or matching placebo
  Interventions: Drug: IMM-BCP-01; Drug: Placebo
- IV Cohort 2 (Experimental): Single intravenous (IV) dose 2 of IMM-BCP-01 or matching placebo
  Interventions: Drug: IMM-BCP-01; Drug: Placebo
- IV Cohort 3 (Experimental): Single intravenous (IV) dose 1 of IMM-BCP-01 or matching placebo
  Interventions: Drug: IMM-BCP-01; Drug: Placebo
- IV Cohort 4 (optional) (Experimental): Single intravenous (IV) dose 4 of IMM-BCP-01 or matching placebo
  Interventions: Drug: IMM-BCP-01; Drug: Placebo

INTERVENTIONS:
Drug: IMM-BCP-01 — Single dose of IMM-BCP-01
Drug: Placebo — Placebo matching single dose of IMM-BCP-01

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of intravenous (IV) IMM-BCP-01 in subjects with mild to moderate COVID-19 through Day 28.

The secondary objectives of the study are to:

* Determine pharmacokinetics (PK) and evaluate viral clearance after single ascending doses of IV IMM-BCP-01 in subjects with mild to moderate COVID-19 through Day 28.
* Evaluate the safety and tolerability, determine PK, and evaluate viral clearance of single ascending doses of IV IMM-BCP-01 in subjects with mild to moderate COVID-19 through Week 12.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 1 study to evaluate the safety, PK, and viral clearance of single ascending doses of IV IMM-BCP-01 in subjects with mild to moderate COVID-19 caused by infection with SARS-CoV-2 and/or its variants.

The study will consist of a screening period of up to 36 hours, a treatment period of one day, two further clinic visits, four visits that will take place either in the clinic or at the subject's home, six virtual visits (telephone or video), and an end-of-study visit 12 weeks (+/- 5 days) after study drug dosing. The total duration of a subject's participation is approximately 90 days.

Subjects presenting at the clinic with signs and symptoms of mild to moderate COVID-19 and agreeing to participate in the study will be screened, and if deemed eligible for the study, will be randomized (2:1) to receive a single IV dose of IMM-BCP-01 or placebo on Day 1. Subjects at risk of severe disease and those who have been vaccinated against COVID-19 within 6 weeks prior to screening or who have received monoclonal antibodies against SARS-CoV-2 and/or COVID-19 convalescent plasma at any time will not be eligible.

Subjects will be randomized to receive IMM BCP-01 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 50 years of age, inclusive, at the time of signing the informed consent.
2. Subjects must have mild to moderate COVID-19 with symptom onset within 5 days prior to study drug administration (see Appendix 13.1 for Food and Drug Administration [FDA] severity guidance). Subjects whose symptoms began >5 days (i.e. ˃120 hours) prior to dosing or whose time of symptom onset cannot be accurately assessed are not eligible.
3. Subjects must have at least 2 of the following COVID-19 symptoms: fever, cough, sore throat, rhinorrhea, malaise, headache, muscle pain, nausea, vomiting, diarrhea, and loss of taste or smell, or other symptoms that the Principal Investigator judges to be referrable to COVID-19.
4. Subjects must be able to maintain oxygen saturation (SpO2) ≥ 94% on room air (no supplemental oxygen).
5. Body mass index ≥ 18.0 and ≤ 30.0 kg/m2.
6. Body weight ≥ 40 kg at screening.
7. Sexually active subjects of reproductive potential must agree to use highly effective contraception from signing of the informed consent through 90 days after infusion of the study drug (see Section 7.4).
8. Males must agree not to donate sperm from dosing until 90 days after administration of the study drug.
9. Subjects must have been in generally good health, as judged by the Principal Investigator, prior to onset of current COVID-19 illness, with no clinically significant medical history.
10. Subjects must be without clinically significant abnormalities as assessed by review of medical and surgical history, physical examination, vital signs measurement, ECG, and laboratory evaluations conducted at screening.

Exclusion Criteria:

1. Has one or more symptoms suggestive of more severe illness with COVID-19 and/or requires hospitalization.
2. Is asymptomatic at screening or randomization, regardless of a positive COVID-19 test.
3. Is at increased risk of severe COVID-19 for any reason including but not limited to: cancer (basal cell carcinoma and prostate carcinoma in situ [Gleason ≤ 6] are acceptable), chronic kidney disease, chronic obstructive pulmonary disease, heart condition (congestive heart failure II, III and IV as per New York Heart Association: coronary disease and any other cardiac condition that imposes high risk of developing severe COVID-19), immunocompromised state from solid organ transplant, sickle cell disease, or other condition, autoimmune disease, use of immunosuppressants (including high doses of systemic corticosteroids), type 1 or type 2 diabetes mellitus, current or prior history of smoking or vaping any product, including nicotine or THC.
4. Has any active infection, other than the underlying COVID-19.
5. Has been admitted to a hospital within 3 months prior to randomization (except for planned admissions for minor procedures).
6. Has been hospitalized due to COVID-19 at any time.
7. Has participated or is participating in a clinical research study currently or within 3 months or less than 5 half-lives of the investigational product (whichever is longer) prior to the screening visit.
8. Has received monoclonal antibodies against SARS-CoV-2 and/or COVID-19 convalescent plasma.
9. Is anticipated to be treated with any approved or investigational drug or agent against SARS-CoV-2 (other than the study drug) during the study including antiviral drug(s), antibodies, or convalescent plasma.
10. Has received any COVID-19 directed treatment in the 3 months prior to the screening visit including but not limited to: Intravenous immunoglobulin, Approved drugs or products used off label for treatment of COVID-19, Other experimental interventions.
11. Has received a COVID-19 vaccination within 6 weeks of screening. Subjects vaccinated ≥ 6 weeks prior to screening and who otherwise meet inclusion/exclusion criteria are eligible to participate.
12. History or suspicion of excessive alcohol use (defined as drinking on average 14 drinks a week for males and 7 drinks a week for females) or of binge drinking (defined as 4 drinks on any day for males and 3 drinks on any day for females, for 5 or more days in the past month)
13. History of substance abuse or current use of any drugs of abuse
14. Any other condition or prior therapy which the Principal Investigator feels may jeopardize the safety of the subject or the objectives of the study.

Note: Other protocol defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) | Up to 28 days
  TEAEs include clinical laboratory values, standard 12-lead ECGs, vital signs, pulse oximetry

SECONDARY OUTCOMES:
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) | Up to 12 weeks
  TEAEs include clinical laboratory values, standard 12-lead ECGs, vital signs, pulse oximetry
PK parameters | Up to 28 days
  measured by maximum observed concentration
PK parameters | Up to 12 weeks
  measured by time to maximum observed concentration
PK parameters | Up to 12 weeks
  measured by terminal elimination half-life
PK parameters | Up to 12 weeks
  measured by clearance
PK parameters | Up to 12 weeks
  measured by volume of distribution
Anti drug antibody | Up to 28 days
  change from baseline
Anti drug antibody | Up to 12 weeks
  change from baseline
Viral clearance | Up to 28 days
  change from baseline
Viral clearance | Up to 12 weeks
  change from baseline

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ark Clinical Research, Long Beach, California
  - Panax Clinical Research, Miami Lakes, Florida
  - Icahn School of Medicine at Mt. Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No